CLINICAL TRIAL: NCT00774124
Title: Improving Outcomes in Underserved Women With GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 071694; 1R21DK071694 (NIH)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus; Pregnancy
Keywords: GDM, pregnancy, macrosomia
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Telemedicine (Experimental): Usual care plus telemonitoring
  Interventions: Other: telemonitoring
- 2 Standard of Care (Active Comparator): Standard of care - women will monitor and record blood glucose levels four times a day.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: telemonitoring — Women will transmit their blood glucose levels, fetal movement counts, and insulin doses via the Internet and/or IVR system at least three times per week
  Arms: 1 Telemedicine
Other: Standard of care — Health data (blood glucose levels and insulin doses) will be recorded in a paper log book which will be reviewed at prenatal visits.
  Arms: 2 Standard of Care

SUMMARY:
Our objective is to test an innovative approach to improve outcomes among underserved women with gestational diabetes. We ill utilize a multi-lingual, Interactive Voice Response (IVR) -enabled telephone system to facilitate diabetes control and thereby improve pregnancy outcomes. Our hypothesis is that Telemonitoring will improve maternal glycemia, thereby reducing infant birth weights and leading to improved pregnancy outcomes.

DETAILED DESCRIPTION:
Using a step care design, women will be randomized into standard of care or Telemonitoring. In the standard of care group, women will monitor their blood glucose levels four times a day, perform fetal movement counting three times a day and also record insulin doses. The women will record this information in a logbook, which will be reviewed by the medical team at prenatal visits. In the Telemonitoring group, women will receive the standard of care anmd will also transmit their blood glucose and fetal movement information to their health care providers.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GDM
* 33 or less weeks gestation

Exclusion Criteria:

* multiple gestations
* history of glucose intolerance outside of pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2007-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
maternal blood glucose control | 3 to 9 months

SECONDARY OUTCOMES:
infant birthweight | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Homko, RN, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Tallahassee Memorial Diabetes Center, Tallahassee, Florida
  - Temple University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Homko CJ, Santamore WP, Whiteman V, Bower M, Berger P, Geifman-Holtzman O, Bove AA. Use of an internet-based telemedicine system to manage underserved women with gestational diabetes mellitus. Diabetes Technol Ther. 2007 Jun;9(3):297-306. doi: 10.1089/dia.2006.0034. PMID 17561800